CLINICAL TRIAL: NCT05920915
Title: The Effect of Cold Application to the Lateral Neck Region on Venous Cannulation Pain: A Prospective Randomized Controlled Study
Brief Title: The Effect of the Cold Application on Venous Cannulation Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Senay Canikli, medical specialist (Anesthesiology and Reanimation), Samsun University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SÜEK-2023 11/19
Record Dates: First submitted 2023-06-08; First posted 2023-06-27 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Venous Cannulation Pain; Nervous Vagus; Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Randomization will be done by closed envelope method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group K (Placebo Comparator): Group K: Control group; 30 seconds (sec) will be waited before the vascular access is opened, no additional action will be taken.
  Interventions: Other: non-interventional clinical research
- Group M (Experimental): Group M: Cold application group; Just before the vascular access was opened, a marble plaque was placed on the carotid (2-3 cm above the clavicle, on the sternocleidomastoid muscle (SCM) 2-3 cm above the clavicle) in the bilateral neck region, 4x5 cm in size, for 30 seconds.
  Interventions: Other: non-interventional clinical research
- Group S (Sham Comparator): Group S: Sham group; Before the vascular access is opened, a marble plaque of 4x5 cm with a polar sheath on it will be applied bilaterally to the neck region of the patients for 30 seconds.
  Interventions: Other: non-interventional clinical research

INTERVENTIONS:
Other: non-interventional clinical research — This study is a non-invasive clinical trial designed to observe the effect of applying cold to the neck area to effect of venous cannulation pain

SUMMARY:
Intravenous (iv) cannulation is one of the most common practices performed by anesthesiologists in and outside the operating room. Vascular access is required before any anesthetic procedure. Venous cannulation is a moderately painful procedure and is uncomfortable for patients, and the pain of intravenous cannulation can increase the patient's stress. Various methods are used to reduce cannulation pain. N. Vagus stimulation is among these methods (1). In this study, we aim to evaluate vascular access pain by stimulating the Nervus Vagus with the cold application method to the neck region of our patients who applied venous cannulation from the back of the hand before anesthesia.

DETAILED DESCRIPTION:
Various ways have been tried to reduce cannulation pain. Methods such as local anesthetic injection to the intervention area, topical anesthetic use, ice application, and vibrating buzzi application were used to relieve the patient's pain and distract him. There are many different methods of stimulating the vagus nerve. The Valsalva maneuver is a mechanism that stimulates the Nervus Vagus (N. Vagus). Stimulation of the vagus nerve is thought to have an analgesic effect (2). Stimulation of the vagal nerve has an antinociceptive effect by triggering the baroreceptor reflex arc. It is thought that a P-like substance is released from the antinociceptive substance with the activation of the baroreceptor reflex arc. The regions where the N. Vagus is most superficial in the periphery are the inner auricle and the lateral neck region. It is also known that cold application to the lateral neck region stimulates the N. Vagus and reduces the heart rate (3). Applying cold to the neck area will have an antinociceptive effect by activating the baroreceptor reflex arc by stimulating the N. vagus. Patients between the ages of 18-70 who will be operated on electively (excluding those who will undergo oncological surgery and those who will undergo cesarean section) will be included in the study. These patients will be evaluated in the anesthesia polyclinic before the operation. Those with scars on the dorsum of the hand, operated on the dorsum of the hand, psoriasis, peripheral vascular disease, chronic analgesic use, opioid use, steroid use, gabapentin use, a history of substance abuse, peripheral neuropathy, oncological treatment, and limited cooperation patients will not be included in the study. The patients will be divided into 3 groups Group K, Group M, and Group S, with 53 people in each group. (The number of patients in the groups was calculated as α=0.05 and β=0.80 when power analysis was performed. The lottery method will be used for randomization.

Group K: Control group; 30 seconds (sec) will wait before the vascular access is opened, no additional action will be taken.

Group M: Cold application group; Just before the vascular access was opened, a marble plaque was placed on the carotid (2-3 cm above the clavicle, on the sternocleidomastoid muscle (SCM) 2-3 cm above the clavicle) in the bilateral neck region, 4x5 cm in size, for 30 seconds.

Group S: Sham group; Before the vascular access is opened, a marble plaque of 4x5 cm with a polar sheath will be applied bilaterally to the neck area of the patients for 30 seconds.

After the patients are taken to the operating room and monitored, we will use the method suitable for the groups we determined by drawing lots. Heart rate (HR), respiratory rate (RR), and noninvasive blood pressure (NIBB) will be recorded before the intravenous line is opened.HR, RR, and NIBB values will be recorded after the application to the neck area. Then, an 18 gauge (green) intravenous cannula will be inserted at once by the same experienced practitioner on the back of the left hand, and patients will be asked to rate their pain levels between 0-10 according to Numerical Rating Scale (NRS), and this value will be recorded. HR, RR, and NIBB values will also be recorded. Patients who cannot be cannulated at once will be excluded from the study.

The data of the patients will be recorded using the Statistical Package for the Social Sciences (SPSS) 18 program. The relationship between the NRS scores of all three groups and the patients' HR, RR, and NIBB values before cold application, after cold application, and during vascular access will be evaluated. Descriptive statistics, analysis of variance, and chi-square test will be used in the evaluation of the data. Mean±standard deviation and percentiles will be used in descriptive statistics. Results will be evaluated at a 95% confidence interval and significance as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* American Society of Anesthesiologists (ASA) I,II,III patients
* Patients who will have elective surgery

Exclusion Criteria:

* Patients undergoing emergency surgery
* Patients who will undergo oncological surgery
* Pregnant patients
* Patients with scars on the back of the hand
* Those who have been operated on the back of the hand
* Patients with psoriasis Those with peripheral vascular disease
* Patients using chronic analgesics
* Patients using opioids
* Those who use steroids Those who use gabapentin
* Those with a history of substance use Those with peripheral neuropathy
* Patients who have received oncological treatment
* Patients with limited cooperation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2023-06-18 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Venous cannulation pain | 5 minutes before induction of anesthesia
  To evaluate the effect of cold application to the neck area on venous cannulation pain. Pain will be scaled from 0 to 10 on a numerical pain scale.
  To evaluate the effect of cold application to the neck area on venous cannulation
  pain.
Heart rate will be evaluated | 5 minutes before induction of anesthesia
  Changes in heart rate will be evaluated (measured in heart rate/minute) during venous cannulation.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa SÜREN, Study Director — Samsun University
Locations (1):
- Şenay Canikli Adıgüzel, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Kumar S, Gautam SK, Gupta D, Agarwal A, Dhirraj S, Khuba S. The effect of Valsalva maneuver in attenuating skin puncture pain during spinal anesthesia: a randomized controlled trial. Korean J Anesthesiol. 2016 Feb;69(1):27-31. doi: 10.4097/kjae.2016.69.1.27. Epub 2016 Jan 28. PMID 26885298
- [Background] Agarwal A, Sinha PK, Tandon M, Dhiraaj S, Singh U. Evaluating the efficacy of the valsalva maneuver on venous cannulation pain: a prospective, randomized study. Anesth Analg. 2005 Oct;101(4):1230-1232. doi: 10.1213/01.ane.0000167270.15047.49. PMID 16192551
- [Background] Jungmann M, Vencatachellum S, Van Ryckeghem D, Vogele C. Effects of Cold Stimulation on Cardiac-Vagal Activation in Healthy Participants: Randomized Controlled Trial. JMIR Form Res. 2018 Oct 9;2(2):e10257. doi: 10.2196/10257. PMID 30684416